CLINICAL TRIAL: NCT01710839
Title: A Phase IV Open Label Trial of the Safety, Tolerability and Efficacy of 0.5mg Ranibizumab Intravitreal Injections Combined With Wide Field Angiography Guided Panretinal Photocoagulation vs. 0.5mg Ranibizumab Intravitreal Injection Monotherapy in Subjects With Ischemic Central Retinal Vein Occlusion, Hemi Retinal Vein Occlusion, and Branch Retinal Vein Occlusion Who Incompletely Respond to at Least 2 Consecutive Intravitreal Injections in the Past 4 Months.
Brief Title: Widefield Angiography Guided Targeted-retinal Photocoagulation Combined With Anti VEgf Intravitreal Injections for the Treatment of Ischemic Central Retinal Vein Occlusion, Hemi Retinal Vein Occlusion, and Branch Retinal Vein Occlusion
Acronym: WAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles C Wykoff, PhD, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Charles C Wykoff, PhD, MD, Deputy Director of Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12246
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Central Retinal, Hemi Retinal & Brach Retinal Vein Occlusions
Keywords: CRVO; BRVO; HRVO; Macular edema; vein occlusion
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Pan Retinal laser combined with 0.5mg ranibizumab (Experimental): Cohort 1 (n=24), previously treated with at least 2 consecutive or more intravitreal injections of any anti-VEGF agent with persistent or recurrent macular edema will receive 6 loading doses of 0.5 mg ranibizumab followed by PRN treatment with ranibizumab 0.5 mg; after receiving the first loading dose of ranibizumab, the subject will have peripheral targeted-retinal photocoagulation (TRP) based on 200° wide field angiography with possibility of a second session of TRP at M4/M7, if non-perfusion persists based on angiogram.The 200°wide field angiography will indicate areas of peripheral ischemia which will be selectively treated, preserving areas of more perfused retina.
  Interventions: Drug: 0.5mg Ranibizumab; Procedure: Targeted Pan Retinal Photocoagulation
- Ranibizumab 0.5mg (Active Comparator): Cohort 2 (n=6), previously treated with at least 2 consecutive or more intravitreal injections of any anti-VEGF agent with persistent or recurrent macular edema will receive 6 loading doses followed by PRN monthly treatment with ranibizumab 0.5 mg.
  Interventions: Drug: 0.5mg Ranibizumab

INTERVENTIONS:
Drug: 0.5mg Ranibizumab — intravitreal injections
  Other Names: Lucentis
Procedure: Targeted Pan Retinal Photocoagulation — Targeted Pan Retinal Photocoagulation based on wide field angiography
  Other Names: PRP; Pan Retinal Photocoagulation; TRP; Pan Laser
  Arms: Targeted Pan Retinal laser combined with 0.5mg ranibizumab

SUMMARY:
To see if Lucentis 0.5mg combined with Targeted Pan Retinal photocoagulation will decrease the total number of intravitreal injections in a year for ischemic central retinal vein occlusion, hemi-retinal vein occlusions and branch retinal vein occlusions compared to standard of care

DETAILED DESCRIPTION:
The WAVE trial is a phase IV, open label, 12-month trial of intravitreal ranibizumab 0.5 mg in patients (n=30) with ischemic CRVO, HRVO and BRVO who have been previously treated with ranibizumab or any other anti-VEGF intravitreal injection therapy, who are incomplete responders to 2 or more consecutive intravitreal anti-VEGF injections in the past 4 months. Randomization is 1:4, 1=control, ranibizumab only, 4=treatment arm. In total, 6 subjects will be randomized to control and 24 randomized to treatment arm.

Cohort 1- 24 Subjects previously treated Patients will receive 6 doses of ranibizumab 0.5 mg, followed by PRN intravitreal injection of ranibizumab 0.5 mg based on pre-defined retreatment criteria for up to 11 total injections.

Wide field angiography guided peripheral targeted-retinal photocoagulation (TRP), will be divided into 2 sessions if needed, one at the 2 weeks post injection visit and another later at M4/V7, if repeat wide field angiogram indicates areas not sufficiently treated in the first TRP session

Cohort 2- 6 Subjects, previously treated patients will receive 6 doses of ranibizumab 0.5 mg, followed by PRN intravitreal injection of ranibizumab 0.5 mg based on pre-defined retreatment criteria for up to 11 total injections.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Visual acuity between 20/25 and 20/800, ETDRS best corrected visual acuity
* Ability to provide written informed consent and comply with study assessments for the full duration of the study

Patients previously treated with any ITV anti-VEGF:

• With at least 2 consecutive monthly intravitreal injections of anti-VEGF medications with presence of persistent or recurrent macular edema in the past 4 months

Exclusion Criteria:

* IOP over 30 mm Hg
* Any previous retinal laser photocoagulation to the study eye
* Previous intravitreal injection in the study eye of any corticosteroid treatment
* Previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
* Intracapsular cataract extraction
* Any previous radiation treatments to head/neck that the principal or sub investigator feels is clinically relevant
* Inability to assess iris or angle neovascularization (corneal opacity precluding gonioscopy)
* Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
* Significant diabetic retinopathy in the fellow eye (diabetic macular edema, proliferative diabetic retinopathy, or high-risk non-proliferative diabetic retinopathy)
* Participation in another simultaneous medical investigator or trial
* Ocular disorders or concurrent disease in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention, including history of retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., DME, AMD, ocular histoplasmosis, or pathologic myopia)
* Structural damage to the center of the macula in the study eye prior to CRVO, HRVO and BRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
* Vitreomacular traction or clinically significant epiretinal membrane in the study eye evident biomicroscopically or by OCT (vitreomacular attachment OK)
* Infectious blepharitis, keratitis, scleritis, or conjunctivitis (in either eye) or current treatment for serious systemic infection
* Spherical equivalent of the refractive error in the study eye of more than -8 diopters myopia (For patients who have had refractive or cataract surgery in the study eye, preoperative spherical equivalent refractive error of more than -8 diopters myopia is not allowed)
* Uncontrolled Blood pressure: defined as systolic pressure > 180mmHg and/or diastolic pressure of >110 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed by the principal investigator (PI) and/or the sub-investigator.
* History of allergy to humanized antibodies or any component of the ranibizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Wykoff, PhD, MD, Principal Investigator — Retina Consultants Houston
Locations (3):
- United States (3):
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

REFERENCES:
- [Background] Armaly MF. Ocular pressure and visual fields. A ten-year follow-up study. Arch Ophthalmol. 1969 Jan;81(1):25-40. doi: 10.1001/archopht.1969.00990010027005. No abstract available. PMID 5763217
- [Background] Boyd SR, Zachary I, Chakravarthy U, Allen GJ, Wisdom GB, Cree IA, Martin JF, Hykin PG. Correlation of increased vascular endothelial growth factor with neovascularization and permeability in ischemic central vein occlusion. Arch Ophthalmol. 2002 Dec;120(12):1644-50. doi: 10.1001/archopht.120.12.1644. PMID 12470137
- [Background] Brown DM, Campochiaro PA, Singh RP, Li Z, Gray S, Saroj N, Rundle AC, Rubio RG, Murahashi WY; CRUISE Investigators. Ranibizumab for macular edema following central retinal vein occlusion: six-month primary end point results of a phase III study. Ophthalmology. 2010 Jun;117(6):1124-1133.e1. doi: 10.1016/j.ophtha.2010.02.022. Epub 2010 Apr 9. PMID 20381871
- [Background] Campochiaro PA, Brown DM, Awh CC, Lee SY, Gray S, Saroj N, Murahashi WY, Rubio RG. Sustained benefits from ranibizumab for macular edema following central retinal vein occlusion: twelve-month outcomes of a phase III study. Ophthalmology. 2011 Oct;118(10):2041-9. doi: 10.1016/j.ophtha.2011.02.038. Epub 2011 Jun 29. PMID 21715011
- [Background] A randomized clinical trial of early panretinal photocoagulation for ischemic central vein occlusion. The Central Vein Occlusion Study Group N report. Ophthalmology. 1995 Oct;102(10):1434-44. PMID 9097789
- [Background] Natural history and clinical management of central retinal vein occlusion. The Central Vein Occlusion Study Group. Arch Ophthalmol. 1997 Apr;115(4):486-91. doi: 10.1001/archopht.1997.01100150488006. PMID 9109757
- [Background] Christen WG, Glynn RJ, Manson JE, Ajani UA, Buring JE. A prospective study of cigarette smoking and risk of age-related macular degeneration in men. JAMA. 1996 Oct 9;276(14):1147-51. PMID 8827967
- [Background] Conn G, Bayne ML, Soderman DD, Kwok PW, Sullivan KA, Palisi TM, Hope DA, Thomas KA. Amino acid and cDNA sequences of a vascular endothelial cell mitogen that is homologous to platelet-derived growth factor. Proc Natl Acad Sci U S A. 1990 Apr;87(7):2628-32. doi: 10.1073/pnas.87.7.2628. PMID 2320579
- [Background] Connolly DT, Heuvelman DM, Nelson R, Olander JV, Eppley BL, Delfino JJ, Siegel NR, Leimgruber RM, Feder J. Tumor vascular permeability factor stimulates endothelial cell growth and angiogenesis. J Clin Invest. 1989 Nov;84(5):1470-8. doi: 10.1172/JCI114322. PMID 2478587
- [Background] Connolly DT, Olander JV, Heuvelman D, Nelson R, Monsell R, Siegel N, Haymore BL, Leimgruber R, Feder J. Human vascular permeability factor. Isolation from U937 cells. J Biol Chem. 1989 Nov 25;264(33):20017-24. PMID 2584205
- [Background] de Vries C, Escobedo JA, Ueno H, Houck K, Ferrara N, Williams LT. The fms-like tyrosine kinase, a receptor for vascular endothelial growth factor. Science. 1992 Feb 21;255(5047):989-91. doi: 10.1126/science.1312256.
- [Background] Hayreh SS, Klugman MR, Podhajsky P, Kolder HE. Electroretinography in central retinal vein occlusion. Correlation of electroretinographic changes with pupillary abnormalities. Graefes Arch Clin Exp Ophthalmol. 1989;227(6):549-61. doi: 10.1007/BF02169451. PMID 2483144
- [Derived] Fan W, Fleming A, Hemert JV, Wykoff CC, Brown DM, Robertson G, Wang K, Falavarjani KG, Sadda SR, Ip M. RETINAL VASCULAR BED AREA IN EYES WITH RETINAL VEIN OCCLUSION ON ULTRA-WIDEFIELD FLUORESCEIN ANGIOGRAPHY: WAVE Study. Retina. 2022 Oct 1;42(10):1883-1888. doi: 10.1097/IAE.0000000000003549. PMID 35976232
- [Derived] Wykoff CC, Ou WC, Wang R, Brown DM, Cone C, Zamora D, Le RT, Sagong M, Wang K, Sadda SR; WAVE Study Group. Peripheral Laser for Recalcitrant Macular Edema Owing to Retinal Vein Occlusion: The WAVE Trial. Ophthalmology. 2017 Jun;124(6):919-921. doi: 10.1016/j.ophtha.2017.01.049. Epub 2017 Mar 18. No abstract available. PMID 28318636

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Started | 24 | 6
Completed | 23 | 0
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg | Total
Number analyzed (Participants) | 24 | 6 | 30
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [43 to 80] | 63.8 [56 to 77] | 64.1 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 13 | 2 | 15
RVO Subtype [Count of Participants; unit: Participants]
  CRVO | 13 | 4 | 17
  BRVO | 9 | 2 | 11
  HRVO | 2 | 0 | 2
Prior Anti-VEGF Injections [Mean (Full Range); unit: injections] | 10.2 [2 to 34] | 10.0 [2 to 41] | 10.1 [2 to 41]
ETDRS BCVA Letters [Mean (Full Range); unit: ETDRS BCVA Letters] — Visual function of the study eye was assessed using the ETDRS protocol, which is a widely accepted international standard for macular laser photocoagulation treatment. A higher score represents better functioning.
  ETDRS BCVA Letters | 51.7 [7 to 77] | 55.3 [29 to 71] | 52.4 [7 to 77]
Central Retinal Thickness [Mean (Full Range); unit: micrometers] | 525 [224 to 1240] | 471 [272 to 910] | 514 [224 to 1240]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Intravitreal Injections Over a 12 Month Period
Description: Assess the number of intravitreal injections over 12 months.
Time Frame: 12 months
Measure: Mean (Full Range); unit: injections
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 24 | 6
injections | 8.7 [5 to 12] | 9.5 [7 to 12]

2. Primary Outcome: Visual Acuity
Description: Evaluate the mean change from baseline in ETDRS best-corrected visual acuity at 12 months. The ETDRS protocol is a widely accepted international standard for macular laser photocoagulation treatment. A higher score represents better functioning.
Time Frame: 12 month period
Population: 1 patient withdrew from the study before month 12
Measure: Mean (Standard Error); unit: ETDRS BCVA Letters
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 23 | 6
ETDRS BCVA Letters | 14.9 (3.4) | 10.7 (4.4)

3. Secondary Outcome: Retinal Ischemia
Description: Quantify change in area of perfused and ischemic retina.
Time Frame: 12 month period
Population: Analysis of this outcome measure is still in progress. Data will be reported when the analysis is completed.
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Foveal Avascular Zone
Description: Assess change in foveal avascular zone area and largest diameter, measured during the early phase of the angiogram
Time Frame: 12 months
Population: Analysis of this outcome measure is still in progress. Data will be reported when the analysis is completed.
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Adverse Events
Description: Incidence and severity of adverse events (ocular and non-ocular).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 24 | 6
Participants
  Notable Ocular Events | 17 | 2
  Serious Non-Ocular Events | 2 | 0

6. Secondary Outcome: Neovascularization of the Iris, Optic Nerve and Elsewhere
Description: Percent of patients that develop neovascularization of the iris, optic nerve and/or elsewhere.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 24 | 6
percentage of patients | 8.33 | 0

7. Secondary Outcome: Central Foveal Outcome
Description: Mean change in Central Foveal Volume on High Resolution OCT.
Time Frame: 12 months
Population: 1 patient withdrew from the study before month 12
Measure: Mean (Standard Deviation); unit: cubic millimeters
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 23 | 6
cubic millimeters | -0.15 (.21) | -0.15 (.20)

8. Secondary Outcome: Aqueous VEGF Levels
Description: VEGF, other cytokines and ranibizumab levels in aqueous and serum samples at randomization and at the exit or early termination visit.
Time Frame: 12 Months
Population: Analysis of this outcome measure is still in progress. Data will be reported when the analysis is completed.
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Visual Field
Description: Goldman Visual Field changes at 6 and 12 months from baseline. Goldmann perimetry is a method used to map a patient's field of vision (central and peripheral). Changes will be assessed by manual digital quantification of GVF plots.
Time Frame: 6 and 12 Months
Population: Patients who completed GVF testing at baseline, M6, and M12 with adequate fixation and cooperation during testing were included in GVF analyses (n=14)
Measure: Mean (Standard Error); unit: square degrees
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Number analyzed (Participants) | 11 | 3
square degrees
  Month 6 | -1269 (180) | 102 (423)
  Month 12 | -1628 (353) | -1875 (326)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab | Ranibizumab 0.5mg
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/6
Other Adverse Events (participants affected / at risk) | 17/24 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab (N=24) | Ranibizumab 0.5mg (N=6)
Hemorrhoids with rectal bleeding (Vascular disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Pan Retinal Laser Combined With 0.5mg Ranibizumab (N=24) | Ranibizumab 0.5mg (N=6)
Glaucoma suspect (Eye disorders) | 1 (1) | 1 (1)
Cataract progression (Eye disorders) | 3 (3) | 1 (1)
Visual distortion (Eye disorders) | 8 (8) | 0 (0)
Posterior vitreous detachment (Eye disorders) | 3 (3) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No